CLINICAL TRIAL: NCT03441308
Title: "Dare to be Satisfied With Food" - a Group Treatment Method for Sustainable Weight Reduction in Adults With BMI 27-45
Brief Title: "Dare to be Satisfied With Food" - a Group Treatment Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORSS-752611
Record Dates: First submitted 2017-12-18; First posted 2018-02-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Overweight and Obesity
Keywords: Dieting; learning to eat; group treatment
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational method of group treatment (Active Comparator): Educational method of group treatment based on regular meals and food based on Nordic nutrition recommendations. The method has been developed by a district nurse at Ljungby. Ten meetings in groups of 6-8 participants over 6 months. Group meeting number 5 includes short individual consultations. In addition, individual consultation after group meeting 1 and 10.
  Interventions: Behavioral: Educational method of group treatment
- Dietary advice (Placebo Comparator): The control group is offered dietary advice according to the Swedish National Food Agency's guidelines for overweight and obesity (including brochures) at one occasion.
  Interventions: Behavioral: Educational method of group treatment

INTERVENTIONS:
Behavioral: Educational method of group treatment
  Other Names: Dietary advice

SUMMARY:
The concept "Dare to be satisfied with food" is an educational method of group treatment based on regular meals and food based on Nordic nutrition recommendations. The method has been developed by a district nurse at the city of Ljungby, Sweden and has shown permanent weight loss in a limited number of persons who tested the method. It is important to test the method scientifically and in the long term for possible implementation in routine activities in the healthcare sector. Adults with overweight and obesity (BMI 27-45) will be recruited to the study by announcing in newspapers in the counties of Kronoberg and Kalmar and then randomized to intervention group and control group, where the control group receives dietary advice according to the Swedish National Food Agency's guidelines for overweight and obesity (including brochures).

DETAILED DESCRIPTION:
The incidence of obesity among adults in Sweden has more than doubled since the 1980s, and the trend seems to continue according to figures from the Public Health Authority (2013), which showed that of the adult population 35% were overweight and 15% obese. Obesity raises the risk of severe diseases such as cardiovascular disease, type 2 diabetes and some cancers. Arthritis, gallstones and childlessness are also common in obese people. In the field of health care, the views differ as to which dietary advice is best for obese people. Swedish Agency For Health Technology Assessment and Assessment of Social Services (SBU, 2013) review of the overall research shows that several types of dietary advice can lead to weight loss. In the long term, councils were equivalent to weight loss, while in the short term a difference between costs was different. As for beverages, a slight intake of sweet drinks showed a weight loss. For some people low blood sugar can lead to uncontrolled eating and were the gateway to improper eating habits.

The aim is to study the effect of the "Dare to be satisfied with food concept" for weight loss with five years follow-up compared to now recommended short counseling according to the Swedish National Food Agency's recommendations.

Participants in the project will be recruited through advertising I newspapers in the counties of Kronoberg and Kalmar. Anyone who meets the criteria and wishes to attend a telephone interview will receive an information letter together with an informed consent form to return. Thereafter, the persons are randomized to the intervention or control group in blocks of 20. The intervention group is offered 10 meetings in groups of 6-8 participants over 6 months. Group meeting 5 includes a short individual consultation. In addition, individual consultation and sampling after group meeting 1 and 10. The control group is offered dietary advise according to the Swedish Food Authority's guidelines for overweight and obesity (including brochures) on an individual occasion including blood samples at the start and after 6 months. At the first visit, a survey is conducted on questions about background factors, living habits, quality of life, health and disease. Sampling includes length, weight, waist and seat measurements, blood pressure, heart rate, blood samples (blood value, blood lipids, metabolism, long-term sugar, electrolytes and liver and kidney function.Then follow-up once yearly for five years for both groups with surveys and sampling in the same way.

Power calculation: At alpha 0.05 and beta 0.2 (power 0.8) 65 people must be randomized in each group to find a weight difference of at least 5 kg. Considering a drop out of about 1/3, 100 people need to be randomized to each group.

Statistical analysis will be done according to intention to treat with major outcome weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 27-45
* Speaks the Swedish language
* Residents of Kronoberg or Kalmar county

Exclusion Criteria:

* Insulin-treated diabetes
* Severe mental illness
* Severe liver disease
* Severe kidney disease
* Heart failure grade 3-4
* Other serious generalized disease
* Multiple food allergy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Weight loss | From baseline to 5 years
  Weight loss of 5 kg or more

SECONDARY OUTCOMES:
Improved lipid profile | From baseline to 5 years
  Lower fasting lipid profile (triglycerides/cholesterol)
Improved quality of live | From baseline to 5 years
  Measured with standard Visual Analog Scale from 0 to100 based on a numeric Likert scale (0 = "very low quality of life", and 100 = "highest possible quality of life"), i.e. Higher scores indicate higher quality of life.
Blood pressure reduction | From baseline to 5 years
  Systolic and diastolic blood pressure
Body fat percentages reduction | From baseline to 5 years
  Body fat percentages measured by bioelectrical impedance analysis (BIA)
Urate reduction | From baseline to 5 years
  Lower urate level

CONTACTS AND LOCATIONS:
Overall Officials: Lena Lendahls, PhD, Study Director — Kronoberg County Council; Sara Holmberg, MD, PhD, Principal Investigator — Kronoberg County Council; Kjell-Ake I Alle, MD, PhD, Principal Investigator — Kronoberg County Council; Mari Bergenholz-Liljedal, Nurse, Study Director — Kronoberg County Council

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data för all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data vill be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by our study group. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Holm S. Obesity interventions and ethics. Obes Rev. 2007 Mar;8 Suppl 1:207-10. doi: 10.1111/j.1467-789X.2007.00343.x. No abstract available. PMID 17316327
- [Background] Karnehed N, Rasmussen F, Hemmingsson T, Tynelius P. Obesity and attained education: cohort study of more than 700,000 Swedish men. Obesity (Silver Spring). 2006 Aug;14(8):1421-8. doi: 10.1038/oby.2006.161. PMID 16988085
- [Background] Lewis S, Thomas SL, Blood RW, Castle DJ, Hyde J, Komesaroff PA. How do obese individuals perceive and respond to the different types of obesity stigma that they encounter in their daily lives? A qualitative study. Soc Sci Med. 2011 Nov;73(9):1349-56. doi: 10.1016/j.socscimed.2011.08.021. Epub 2011 Sep 10. PMID 21944718
- [Background] Zhang C, Rexrode KM, van Dam RM, Li TY, Hu FB. Abdominal obesity and the risk of all-cause, cardiovascular, and cancer mortality: sixteen years of follow-up in US women. Circulation. 2008 Apr 1;117(13):1658-67. doi: 10.1161/CIRCULATIONAHA.107.739714. Epub 2008 Mar 24. PMID 18362231
- [Background] Nygardh A, Malm D, Wikby K, Ahlstrom G. The experience of empowerment in the patient-staff encounter: the patient's perspective. J Clin Nurs. 2012 Mar;21(5-6):897-904. doi: 10.1111/j.1365-2702.2011.03901.x. Epub 2011 Nov 15. PMID 22081948
- See also: The Public Health Agency of Sweden (2017). National Public Health Data:overweight and adiposity.[2017-02-26] — http://www.folkhalsomyndigheten.se
- See also: New Nordic Nutrition Recommendations are here. Food & Nutrition Research — http://dx.doi.org/10.3402/fnr.v57i0.22903
- See also: Swedish Council on Health Technology Assessment.Food with adiposity: a systematic literature review (SBU report) [2013] — http://www.sbu.se